CLINICAL TRIAL: NCT04820582
Title: Defining a Standard Set of Value-Based Patient-Centered Outcomes for Endometriosis: A Delphi Study Conducted by the Study Group VALue Based HEalth CaRe In Endometriosis (VALHERIE).
Brief Title: Defining a Standard Set of Value-Based Patient-Centered Outcomes for Endometriosis
Status: Completed | Type: Observational
Sponsor: One Clinic (Other)
Collaborators: Poissy-Saint Germain Hospital (Other); Versailles Saint-Quentin-en-Yvelines University (Other); PointGyn (Unknown)
Responsible Party: Sponsor
Other Study IDs: Endo001
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Endometriosis
Keywords: Endometriosis; Delphi Study; Patient Reported Outcome Measures (PROMs); Clinician Reported Outcome Measures (CROMs)
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi Panel: A group of international experts comprising patients experts, gynecologists, radiologist, psychologists, nurses and researchers, were identified based on their expertise in the field or due to your active role in an endometriosis patient association that have accepted to participate to this study.
  Interventions: Other: Delphi Questionnaire

INTERVENTIONS:
Other: Delphi Questionnaire — Evaluation of a list of PROMs and CROMs specific for endometriosis (previously selected from a litterature review) on a Likert scale of 1 to 9 for their relevance and feasibility

SUMMARY:
Endometriosis is a chronic disease that affects one out of 10 women. Endometriosis care is full of variation. Recommendations for optimal management vary between clinician and centers. One way of dealing with this unwanted variation is the shift towards a value -based endometriosis care. Value-based healthcare (VBHC) is a strategy focused on the optimization of the balance between outcomes that are important to patients and cost to achieve these outcomes. To do so, for a given condition it is important to define a standardized set of outcomes metrics allowing quality of care monitoring and comparison in order to optimize clinical practices and patient pathways. A common set of outcomes combining clinical outcomes (Clinical Reported Outcome Measures, CROMs) as well as quality of life and functional recovery indicators through Patient Reported Outcome Measures (PROMs). Different standardized data sets have already been developed to measure outcomes in other pathologies, however a standardized set of outcome measurements have not yet been determined for endometriosis. The objective of this study is to determine a standard set of outcome measurements for endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Profession: gynecologists, radiologist, psychologists, nurses and researchers having an expertise in the field of endometriosis
* Patient experts having an active role in an endometriosis patient association

Exclusion Criteria:

* Retirement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A group of international experts comprising patients experts, gynecologists, radiologist, psychologists, nurses and researchers, that have been identified based on their expertise in the field or due to their active role in an endometriosis patient association
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Agreement on a list of PROMs and CROMs that are relevant and feasible in endometriosis care by the expert panel | 6 months
  Agreement is defined as a consensus of 70% between expert panel members

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Intercomunal Poissy Saint Germain en Laye, Poissy, France

IPD SHARING:
Plan to Share IPD: No